CLINICAL TRIAL: NCT01897298
Title: Effectiveness of an Intervention of Urban Training in Patients With Chronic Obstructive Pulmonary Disease (COPD): a Randomised Controlled Trial
Brief Title: Urban Training for COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Judith Garcia-Aymerich (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Sociedad Española de Neumología (SEPAR), Barcelona (Unknown); University Ramon Llull (Other); Hospital Clinic of Barcelona (Other); Hospital del Mar (Other); Germans Trias i Pujol Hospital (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Hospital de Mataró, Mataró (Unknown); Hospital de Viladecans, Viladecans (Unknown); Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor-Investigator, Judith Garcia-Aymerich, Associate Research Professor, Barcelona Institute for Global Health
Organization: Barcelona Institute for Global Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI11/01283; 147/2011 (Other Grant/Funding Number: SEPAR)
Record Dates: First submitted 2013-07-03; First posted 2013-07-11 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: chronic obstructive pulmonary disease (COPD); urban training; physical activity; active aging
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Urban training Intervention (Experimental): Patients will be advised to walk in the defined urban trails.
  Interventions: Behavioral: Urban training
- Usual care (No Intervention): Patients will continue their usual care

INTERVENTIONS:
Behavioral: Urban training — Recommendation to walk a minimum of 5 days per week in urban walkable trails appropriate for the patient.
  Arms: Urban training Intervention

SUMMARY:
This project plans on a training intervention by using public spaces and urban walkable trails, adapted to each patient needs and capabilities. Primary objective is to assess 12 months effectiveness of the intervention with respect to: (primary outcome): physical activity level, and (secondary outcomes): COPD admissions, exercise capacity, body composition, quality of life, and mental health.

ELIGIBILITY:
Inclusion Criteria:

* age > 45 years
* COPD diagnosed by pulmonary function tests during clinical stability, with a ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) ≤ 0.70
* clinical stability, defined as at least 4 weeks without antibiotics or oral corticosteroids.

Exclusion Criteria:

* living >6 months/year outside of the included municipalities,
* living to a distance higher than 500 meters to any of the urban trails used for the study,
* mental disability according to the Mini Mental State Examination in its validated Spanish version
* comorbidity that could interfere with study tests (e.g., lower limb amputation)
* severe psychiatric disease or severe comorbidity limiting survival at one year, according to medical history.

Ages: 45 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2013-07; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Baseline and 12 months follow-up
  Change in physical activity between baseline and 12 months follow-up, as defined by average steps per day measured with an activity monitor

SECONDARY OUTCOMES:
COPD admissions to emergency-room or hospital | 12 months follow-up
Change in exercise capacity, as measured with 6-min walking distance | Baseline and 12 months
  Change in exercise capacity between baseline and 12 months, as measured with 6-min walking distance
Change in body weight and composition | Baseline and 12 month
  Change in body weight and composition between baseline and 12m follow-up, as measured with bioimpedance
Change in quality of life | Baseline and 12-m
  Change in quality of life between baseline and 12-m follow-up, as measured with CAT and CCQ
Change in anxiety and depression symptoms | Baseline and 12 months
  Change in anxiety and depression symptoms between baseline and 12 months follw-up, as measured with the HAD scale

OTHER OUTCOMES:
Changes in cognitive status | Baseline and 12months
  Changes between baseline and 12 months follow-up in cognitive status measured with the Phototest
Changes in the Clinical PPAC | Baseline and 12months
  Changes between baseline and 12 months follow-up in phsyical activity measured with the Clinical visit "PROactive Physical Activity in COPD" instrument

CONTACTS AND LOCATIONS:
Overall Officials: Judith Garcia-Aymerich, MD PhD, Principal Investigator — Centre for Research in Environmental Epidemiology (CREAL)
Locations (5):
- Spain (5):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - CAP Maresme, Mataró, Barcelona
  - CAP Maria Bernades, Viladecans, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Clinic, Barcelona

REFERENCES:
- [Derived] Delgado-Ortiz L, Arbillaga-Etxarri A, Rodriguez-Chiaradia DA, Gimeno-Santos E, Barberan-Garcia A, Balcells E, Rodriguez-Roisin R, Garcia-Aymerich J. Physical activity and cardiac autonomic dysfunction in patients with chronic obstructive pulmonary disease: A cross-sectional analysis. Ann Phys Rehabil Med. 2022 May;65(3):101501. doi: 10.1016/j.rehab.2021.101501. Epub 2021 Nov 22. PMID 33662597
- [Derived] Koreny M, Demeyer H, Arbillaga-Etxarri A, Gimeno-Santos E, Barberan-Garcia A, Benet M, Balcells E, Borrell E, Marin A, Rodriguez Chiaradia DA, Vall-Casas P, Vilaro J, Rodriguez-Roisin R, Garcia-Aymerich J. Determinants of study completion and response to a 12-month behavioral physical activity intervention in chronic obstructive pulmonary disease: A cohort study. PLoS One. 2019 May 20;14(5):e0217157. doi: 10.1371/journal.pone.0217157. eCollection 2019. PMID 31107900
- [Derived] Arbillaga-Etxarri A, Gimeno-Santos E, Barberan-Garcia A, Balcells E, Benet M, Borrell E, Celorrio N, Delgado A, Jane C, Marin A, Martin-Cantera C, Monteagudo M, Montella N, Munoz L, Ortega P, Rodriguez DA, Rodriguez-Roisin R, Simonet P, Toran-Monserrat P, Torrent-Pallicer J, Vall-Casas P, Vilaro J, Garcia-Aymerich J. Long-term efficacy and effectiveness of a behavioural and community-based exercise intervention (Urban Training) to increase physical activity in patients with COPD: a randomised controlled trial. Eur Respir J. 2018 Oct 18;52(4):1800063. doi: 10.1183/13993003.00063-2018. Print 2018 Oct. PMID 30166322
- [Derived] Arbillaga-Etxarri A, Gimeno-Santos E, Barberan-Garcia A, Benet M, Borrell E, Dadvand P, Foraster M, Marin A, Monteagudo M, Rodriguez-Roisin R, Vall-Casas P, Vilaro J, Garcia-Aymerich J; Urban Training Study Group. Socio-environmental correlates of physical activity in patients with chronic obstructive pulmonary disease (COPD). Thorax. 2017 Sep;72(9):796-802. doi: 10.1136/thoraxjnl-2016-209209. Epub 2017 Mar 1. PMID 28250201